CLINICAL TRIAL: NCT06864000
Title: Phenotypic and Molecular Characterisation of Early-onset Cerebral Amyloid Angiopathy
Brief Title: Phenotypic and Molecular Characterisation of Cerebral Amyloid Angiopathy
Acronym: GENERALITY2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0241/OB; 2022-A02248-35 (Other: French Minister)
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Amyloid Aβ Angiopathy
Keywords: Phenotypic and molecular characterisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Study of the enrichment of rare and pathogenic variants in candidate genes such as APOE, SORL1, TREM2, ABCA7, ABCA1 and ATP8B4 and possibly new genes in a population of Aβ-AAC patients compared with a cohort population of healthy FREX volunteers (via genetic association testing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FREX (French Exome Project) control cohort group: Control cohort corresponding to the FREX cohort (French Exome Project) including 585 exomes of healthy individuals (from 6 French regions) and whose data is already available to research groups for case-control association analysis.
- Group of patients with cerebral amyloid angiopathy (CAA): Patients with APOE4 genetic risk factors and rare variants of SORL1, TREM2, ABCA7, ABCA1 and ATP8B4

SUMMARY:
Cerebral Aβ amyloid angiopathy is a severe disease characterised by amyloid deposits in the cerebral vessels, manifested mainly by recurrent cerebral haematomas and cognitive impairment. Diagnostic criteria are based on brain imaging, but the usefulness of this imaging in predicting the course of the disease remains undetermined. The genetic component is largely understudied. Less than 5% of patients carry mutations or duplications of the APP gene. Susceptibility factors such as APOE genotypes and rare variants recently discovered in Alzheimer's disease within the SORL1, TREM2 or ABCA7, ABCA1 and ATP8B4 genes could play a role in the pathophysiology of cerebral amyloid angiopathy. There is currently no specific treatment available. Based on a national recruitment of patients with cerebral amyloid angiopathy, this project aims to assess the role of genetic variants in the diagnosis and progression of cerebral amyloid angiopathy. A better understanding of the mechanisms, particularly genetic, could help us to develop treatments in the era of gene therapy.

DETAILED DESCRIPTION:
This research is carried out on the same blood sample taken during the treatment and sent to the Rouen University Hospital Genetics Laboratory for research into point mutations or duplication of the APP gene as part of the diagnosis of cerebral amyloid angiopathy (CAA). For each gene, the proportions of variant carriers will be compared between cases and controls using a Fisher exact test with R statistical software. To rule out any population stratification bias, the tests will also be carried out using logistic regression adjusted on the first PCA axes (principal component analysis) using the seqmeta function. A Bonferroni correction will then be used to adjust the significance threshold according to the number of genes tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cerebral amyloid angiopathy (CAA) whose genetic samples are initially sent to the Rouen or Paris-Lariboisière genetics laboratories for molecular diagnosis of a genetic cause, thanks to national recruitment and for whom the patients consent to continuing genetic analyses for research purposes without feedback.
* Diagnosis of cerebral amyloid angiopathy (CAA) certain or probable according to the modified Boston diagnostic criteria (1) (except age)
* Age of onset of symptoms <66 years
* Absence of APP mutation/duplication (analysis must already have been carried out in the laboratory on receipt of the sample as part of routine care)
* Signed consent for research
* Patient covered by a social security scheme

Exclusion Criteria:

* Age at first neurological symptom > 66 years
* Minor patients
* Other differential diagnosis that better explains the clinical situation
* Identification of mutations or duplication of the APP gene
* AAC possible but not probable according to the revised Boston criteria
* Patient deprived of liberty by judicial or administrative decision

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Etude proposée aux patients adultes atteints d'angiopathie amyloïde cérébrale pour lesquels un prélèvement sanguin est prévu au titre du diagnostic dans le cadre du soin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
patients with APOE4 genetic risk factors | 1 day
  Define the proportion of patients with APOE4 genetic risk factors (%) in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.
patients with rare variants of SORL1 | 1 day
  Define the proportion of patients with rare variants (%) of SORL1, in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.
patients with rare variants of TREM2 | 1 day
  Define the proportion of patients with rare variants (%) of TREM2 in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.
patients with rare variants of ABCA7 | 1 day
  Define the proportion of patients with rare variants (%) of ABCA7 in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.
patients with rare variants of ABCA1 | 1 day
  Define the proportion of patients with rare variants (%) of ABCA1 in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.
patients with rare variants of ATP8B4 | 1 day
  Define the proportion of patients with rare variants (%) of ATP8B4 in patients with early-onset cerebral amyloid angiopathy (CAA) (<66 years) and patients with causal mutations in the PSEN1 and PSEN2 genes.

SECONDARY OUTCOMES:
Genotype/clinical phenotype correlations | 12 months
  Establish genotype/clinical phenotype correlations concerning the age of onset, the severity of the disease and the risk of recurrence of haematomas (identified during follow-up visits at M6 and M12 as part of routine care).
Biological characterisation of AACs (Aβ42,CSF biomarkers) | 12 months
  - assessment of the diagnostic value of assays for Aβ42 biomarkers currently validated in Alzheimer's disease and related neurocognitive disorders
Biological characterisation of AACs (Aβ40, CSF biomarkers) | 12 months
  - assessment of the diagnostic value of assays for Aβ40, CSF biomarkers currently validated in Alzheimer's disease and related neurocognitive disorders
Imaging characterisation of AACs (topography of cerebral bleeds) | 12 months
  - identification of biomarker profiles linked to the topography of cerebral bleeds
Imaging characterisation of AACs (typology of cerebral bleeds) | 12 months
  - identification of biomarker profiles linked to the typology of cerebral bleeds
Imaging characterisation of AACs (distribution of cerebral bleeds) | 12 months
  - identification of biomarker profiles linked to the distribution of cerebral bleeds

CONTACTS AND LOCATIONS:
Overall Officials: Lou LG GRANGEON, Doctor, Principal Investigator — University Rouen Hospital
Locations (1):
- University Hospital Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.